CLINICAL TRIAL: NCT00798278
Title: Exploratory Multicentre Clinical Trial to Compare the Efficacy of Urokinase Versus Video-assisted Thoracoscopic for Treatment of Complicated Parapneumonic Empyema in Childhood
Brief Title: Urokinase Versus Video-assisted Thoracoscopic to Treat Complicated Parapneumonic Empyema in Childhood
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Society of Pediatric Surgery (Other)
Responsible Party: Claudia Marhuenda Irastorza, University Hospital Vall d'Hebron. Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKVATS2007; EudraCT Number 2007-003416-61
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2008-11

CONDITIONS: Empyema; Pneumonia
Keywords: Empyema; Urokinase; Thoracoscopic; Childhood
MeSH Terms: conditions — Empyema; Pneumonia | interventions — Urokinase-Type Plasminogen Activator; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urokinase (Experimental): urokinase infusion for 3 days
  Interventions: Drug: Urokinase
- Thoracoscopic (Active Comparator): Video-Assisted Thoracoscopic
  Interventions: Procedure: Video-Assisted Thoracoscopic

INTERVENTIONS:
Drug: Urokinase — Chest tube with intrapleural urokinase infusion for 3 days
  Arms: Urokinase
Procedure: Video-Assisted Thoracoscopic — Video-Assisted Thoracoscopic decortication
  Arms: Thoracoscopic

SUMMARY:
A great controversy exists about which is the best method to perform the evacuation of the collection. The purpose of this study is to evaluate which is the best initial treatment to drain complicated parapneumonic empyema (stages II and III) in children: the present study raises a hypothesis of equivalence between both arms of treatment (chest drainage plus intrapleural urokinase or videothoracoscopic debridement).

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 15 years of age with pneumonia and persistent fever, and complicated parapneumonic empyema (septation or loculation seen on ultrasound or Rx thorax)stages II and III requiring an intervention to drain

Exclusion Criteria:

* Existing contraindications or other previous conditions, hypertension, pneumothorax

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
duration of the hospital stay after the treatment | 3 months

SECONDARY OUTCOMES:
complications of the treatment and complications of the disease | 3 months
total duration of the hospital stay | 3 months
number of days carrying the chest drain | 3 months
duration of the fever once the empyema has been drained | 3 months

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - University Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital de Donostia, San Sebastián, Donostia
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Infantil La Paz, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias